CLINICAL TRIAL: NCT03445338
Title: A Multiple Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of K0706 in Plasma and Cerebrospinal Fluid in Healthy Volunteers
Brief Title: To Evaluate the Safety, Tolerability and Pharmacokinetics of K0706 in Plasma and Cerebrospinal Fluid in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLR_17_06
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Drug: K0706
- Cohort 2 (Experimental)
  Interventions: Drug: K0706
- Cohort 3 (Experimental)
  Interventions: Drug: K0706

INTERVENTIONS:
Drug: K0706 — Study
  Arms: Cohort 1
Drug: K0706 — Study
  Arms: Cohort 2
Drug: K0706 — Study
  Arms: Cohort 3

SUMMARY:
This is an open-label, multiple-dose study to evaluate the plasma and CSF pharmacokinetics of K0706 in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male subjects, 18 to 45 years of age, inclusive, at screening.
2. Willing and able to give written, and dated an informed consent.
3. Willing and able to comply with the scheduled visits, treatment plan, laboratory testing, study procedures, and restrictions in the Investigator's opinion, and be accessible for follow-up.
4. Medically healthy on the basis of medical history and physical examination.
5. Subjects enrolled in the study should not father a child and follow the necessary precautionary measure to be taken during the course of the study.

Exclusion Criteria:

1. Subjects with a history of a frequent headache, nausea, or vomiting suggestive of increased intracranial pressure.
2. Subject report of recent (6-month) alcohol abuse or illicit drug use or who tests positive at screening, Check-in, or outpatient Visits for breath alcohol and/or drugs of abuse or cotinine;
3. Subjects with a history of any relevant allergy/hypersensitivity.
4. Subjects determined by the investigator to have any medical condition that could jeopardize their health or prejudice the results.
5. Subjects who have participated in CSF collection studies within 56 days prior to check-in.
6. Subjects who donated plasma within 14 days prior to the check-in visit.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
minimum concentration of study drug cerebrospinal fluid (CSF) | Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC Site 1, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102